CLINICAL TRIAL: NCT03711747
Title: Indications for Osteochondral Allograft Transplantation by Evaluating Safety and Efficacy of Total Biologic Total Joint Replacement of Ankle Post-traumatic Osteoarthritis (PTOA)
Brief Title: Indications for Osteochondral Allograft Transplantation
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, James Stannard, Professor, Orthopedic Surgery, University of Missouri-Columbia
Other Study IDs: 2011144
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Post-Traumatic Osteoarthritis of Ankle; Ankle Osteoarthritis; Ankle Injuries
Keywords: Ankle; Ankle Pain; Joint Pain; Ankle Osteoarthritis
MeSH Terms: conditions — Ankle Injuries; Arthralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-traumatic Ankle OA: Post-traumatic ankle OA and requiring osteochondral allograft to tibia and/or talus in ankle
  Interventions: Procedure: Osteochondral allograft ankle

INTERVENTIONS:
Procedure: Osteochondral allograft ankle — Open osteochondral allograft to replace the cartilage that is grade four on the tibia and/or talus

SUMMARY:
With IRB approval, a prospective single-cohort clinical trial will be performed to assess safety and efficacy of total biologic arthroplasty of the ankle. With informed consent, patients (n=10) who require tibio-talar arthroplasty based on physical examination and diagnostic imaging will be enrolled. Primary criteria for inclusion will be Grade IV changes in the articular cartilage of the tibial plafond and/or talar dome as determined by physical examination, diagnostic imaging and/or arthroscopy by the attending surgeon. Exclusion criteria include acute injury to any other part of the affected lower extremity or inability to comply with the protocol.

After enrollment, patients will undergo standard ankle radiography and complete assessments (described below). Size-matched (standard clinical methodology) MOPSTM allografts (Musculoskeletal Transplant Foundation, Edison, NJ) from the same donor will be obtained to treat the entire tibiotalar joint. The affected joint will be treated with OCA transplants using our current technique and instrumentation. Osteochondral grafts including MOPSTM OCAs are regulated under U.S. Food and Drug Administration (FDA) section 361 of the Public Health Service Act and 21 Code of Federal Regulation 1271 that defines human cells, tissues or cellular or tissue based products (HCT/P).

Patients will follow a managed post-operative rehabilitation protocol that is standard for those that have had an osteochondral allograft to their ankle.

Range of motion and patient-reported outcome measures (PROMs) including VAS pain score, AOFAS, and PROMIS Mobility as well as complete radiographs (XR) of the affected ankle will be obtained prior to surgery and at 6 weeks, 3 months, 6 months, and 12 months after surgery to evaluate healing, function and evidence for arthrosis. MRIs for cartilage composition (12 months after surgery, and serum and urine biomarkers for treatment monitoring (preop, 6 and 12 months after surgery) will be performed. We will document all adverse events and complications, including joint or incision infection, graft failure, hardware failure, and arthrofibrosis. Patients with a VAS pain score >5 beyond 3 months postoperatively or clinical or diagnostic imaging evidence for nonunion or graft collapse will undergo MRI of the ankle to determine the appropriate clinical course of action. OCA survival will be determined based on maintenance of acceptable levels of pain (<2 VAS) and function and/or need for revision surgery or total ankle arthroplasty, fusion, or amputation.

ELIGIBILITY:
Inclusion Criteria:

i. Grade IV changes in the articular cartilage of the tibial plafond and/or talar dome as determined by physical exam, diagnostic imaging, and/or arthroscopy by the attending surgeon ii. Between the age of 18-55

Exclusion Criteria:

i. Acute injury to any other part of the affected lower extremity ii. Inability to comply with protocol iii. BMI greater than 40 iv. The subject is either pregnant or a prisoner v. Currently involved in worker's compensation case at the time of enrollment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: With informed consent, patients (n=10) who require tibio-talar arthroplasty based on physical examination and diagnostic imaging will be enrolled. Primary criteria for inclusion will be Grade IV changes in the articular cartilage of the tibial plafond and/or talar dome as determined by physical examination, diagnostic imaging and/or arthroscopy by the attending surgeon. Exclusion criteria include acute injury to any other part of the affected lower extremity or inability to comply with the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) score | 12 Months
  Pain assessment which measures what a patient rates their pain between 0 and 10, with 0 being no pain, and 10 being the most pain

SECONDARY OUTCOMES:
American Orthopaedic Foot and Ankle Society (AOFAS) score | 12 Months
  This measurement tool measures a patient's function out of 100, with 100 being highest amount of function
PROMIS - Physical Function and Mobility | 12 Months
  A survey related to physical function and mobility

CONTACTS AND LOCATIONS:
Overall Officials: James Stannard, MD, Principal Investigator — University of Missouri, Department of Orthopaedic Surgery
Locations (1):
- Missouri Orthopaedic Institute, Columbia, Missouri, United States